CLINICAL TRIAL: NCT04438395
Title: Dielectric Tissue Imaging in Cavotricuspid Isthmus Ablation
Acronym: ERUCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: EPD Solutions, A Philips Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-00016
Record Dates: First submitted 2020-05-18; First posted 2020-06-18 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation and Flutter
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Enrolled AFL and AF Patients: All subjects that are enrolled are group one, as there is only one group of subjects in this study
  Interventions: Device: Cardiac ablation via catheter

INTERVENTIONS:
Device: Cardiac ablation via catheter — Cardiac ablation with a catheter to treat atrial flutter and/or atrial fibrillation

SUMMARY:
This is a prospective, single center, non-randomized, open-label, single arm study in which we will gather data and physician input for the assessment and further development of the KODEX - EPD functions for assessing tissue pressure, tissue thickness, lesion transmurality.

DETAILED DESCRIPTION:
This is a prospective, single center, non-randomized, open-label, single arm study in which we will gather data and physician input for the assessment and further development of the KODEX - EPD functions for assessing tissue pressure, tissue thickness, lesion transmurality. The study will include up to 30 subjects. We will enroll patients with atrial flutter and patients with atrial fibrillation who are scheduled to undergo RF ablation of the cavotricuspid isthmus (CTI). Both male and female subjects who meet all eligibility criteria and give written informed consent will be enrolled in the study. We will be assessing the feasibility of the KODEX-EPD tissue pressure (TP), tissue thickness and lesion transmurality applications.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be aged >18 years.
2. Subject must have signed a written Informed Consent form to participate in the study, prior to any study related procedures.
3. Subject must be willing to comply with the protocol requirements.
4. A female subject is eligible if not of child bearing potential or has a negative pregnancy test within the previous 7 days.
5. Subject is deemed amenable to therapeutic ablation for atrial flutter or atrial fibrillation.

Exclusion Criteria:

1. Any planned surgical or endovascular intervention within 30 days before or after the index procedure.
2. Subject is enrolled in another drug or device study protocol that has not reached its primary endpoint.
3. Patient had experienced previous stroke (TIA or CVA).
4. Thrombi detected in the heart.
5. Known marked valvular insufficiency (moderate-severe and severe)
6. Life expectancy less than 12 months.
7. Known severe renal insufficiency (stages G4 and G5, characterized by severe reduction in GFR [15-29 ml/min/1.73 m2] and GFR [<15 ml/min/1.73 m2], respectively).
8. Subjects that according to the clinical judgment of the caring physician do not fit for the study.
9. Previous right atrial ablation procedure or cardiac ablation procedure performed within 90 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Atrial Flutter and patients with Atrial Fibrillation scheduled to undergo RF ablation of the cavotricuspid isthmus (CTI). Both male and female subjects who meet all eligibility criteria and give written informed consent will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The feasibility of KODEX-EPD tissue pressure (TP) application | During procedure
  • will be evaluated based on comparison with qualitative assessment of catheter contact by the physician during the procedure. We will ask the physician to estimate the level of pressure applied by categorizing the pressure as: no touch, touch (light), touch (firm), or high touch.
The feasibility of KODEX-EPD tissue thickness application | During procedure
  * thickness values will be evaluated by checking whether they are in the range of what can be expected based on feedback from the physician upon review after the treatment (measured in mm)
  * reproducibility of thickness assessment with KODEX-EPD will be calculated from repeat assessments of the same line (measured in mm)
  * relative thickness values will be compared against relative thickness values measured with ICE (measured in mm)
  * relative thickness values will be compared against relative thickness values derived from pre-procedural CT (measured in mm)
The feasibility of KODEX-EPD lesion transmurality application | During procedure
  • will be evaluated by checking whether assessments are reasonable from what can be expected based on feedback from the physician upon review after the treatment. The physician's response will be recorded as yes or no for transmurality.

CONTACTS AND LOCATIONS:
Overall Officials: Larry Chinitz, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States